CLINICAL TRIAL: NCT05122624
Title: PredicTB: Validating a Clinical Risk Score for Early Management of Tuberculosis in Ugandan Primary Health Clinics
Brief Title: A Clinical Risk Score for Early Management of TB in Uganda
Acronym: PredicTB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: R21AI161301 (NIH); R21AI161301 (NIH); IRB00015699 (Other: JHSPH IRB)
Record Dates: First submitted 2021-11-01; First posted 2021-11-17 (Actual); Results first posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-06

CONDITIONS: Tuberculosis, Pulmonary
MeSH Terms: conditions — Tuberculosis, Pulmonary

STUDY DESIGN:
Intervention Model Description: The study includes an intervention arm (four clinics) and a control arm (four clinics).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Score intervention arm (Experimental): The PredicTB score will be implemented in this arm.
  Interventions: Other: PredicTB score
- Control arm (No Intervention): The standard of care will be conducted in this arm.

INTERVENTIONS:
Other: PredicTB score — This is an easy-to-use clinical risk score designed to improve early management of tuberculosis in highly resource-constrained settings where same-day microbiological testing is unavailable. It consists of readily accessible demographic and clinical data and is scored from 1-10.
  We will train clinic staff in eight clinics (four study clinics and four comparison clinics) on the Ugandan standard of care for the diagnosis and treatment of TB. In addition, in the four study clinics, we will provide training on the PredicTB score.
  Arms: Score intervention arm

SUMMARY:
Although curative treatment exists, tuberculosis (TB) remains the leading cause of infectious mortality worldwide - often because people seek care for TB symptoms in highly resource-constrained clinics that cannot provide same-day diagnostic testing. The research team has developed an easy-to-use clinical risk score that, if implemented in these settings, might help clinicians identify patients at high risk for TB and thereby start treatment for those patients on the same day. This study will investigate the effectiveness and implementation of this score in four peri-urban clinics in Uganda, providing critical pragmatic data to inform (or halt) the design of a definitive large-scale cluster randomized trial.

DETAILED DESCRIPTION:
An estimated 1.5 million people die of tuberculosis (TB) every year. Many of these are people who seek care in under-resourced clinics (for example, in rural areas or informal settlements) where same-day TB diagnosis is not available. These patients are often unable to return promptly to receive their results and start treatment, resulting in ongoing disease transmission and often death. If TB treatment could be started on the same day as these patients initially seek care, substantial mortality and transmission could be averted. The research team has developed and validated a clinical risk score ("PredicTB") for adult pulmonary TB that could aid in clinical decision-making. This risk score ranges from 1-10, can be calculated by hand in under a minute using readily available clinical data (e.g., age, sex, self-reported HIV status), and has sufficiently high accuracy to inform decisions about same-day empiric treatment initiation while confirmatory test results are pending. Same-day treatment initiation improves patient outcomes for other infectious diseases (for example, sexually transmitted diseases including HIV), and this novel clinical risk score holds similar promise for TB, the leading cause of infectious mortality worldwide. However, before conducting a large-scale cluster randomized trial to evaluate whether this score could improve patient-important outcomes, it is critical to first generate evidence that this score could be effective and be implemented in the most-resource-limited settings for which it is intended.

The research team proposes a type 2 hybrid effectiveness-implementation evaluation of the PredicTB clinical risk score in four peri-urban clinics in Uganda, with an additional four clinics serving as a comparison group. The Specific Aims are to evaluate the effectiveness of PredicTB on clinical outcomes including rapid treatment initiation, TB mortality, and loss to care (Aim 1); to evaluate the implementation of PredicTB in terms of reach, adoption, implementation, and maintenance (Aim 2); and the project the long-term impact and cost-effectiveness of PredicTB implementation (Aim 3). The primary outcome is the increase in the proportion of patients with microbiologically confirmed TB who start treatment within seven days of initial presentation. To accomplish these aims, the research team will adopt a highly pragmatic study design in which the research team train clinicians in the use of the PredicTB score and perform quarterly site visits but otherwise minimize contact between study staff and treating clinicians. This will enable the research team to evaluate whether implementation of PredicTB is likely to impact clinical decision-making and patient outcomes under actual field settings. If successful, this evaluation will provide critical data to justify (or halt) the conduct of a large-scale pragmatic clinical trial - not only will it generate preliminary evidence of effectiveness, but it will also inform appropriate implementation. Patients in highly resource-constrained settings are at the greatest risk of suffering the ill effects of TB disease, including long-term morbidity and death. This study represents an important first step toward improving clinical management for these marginalized patients and thus toward reaching global targets for ending the TB epidemic.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients submitting sputum for a new diagnosis of pulmonary TB in the four study clinics and four comparison clinics between month -6 and month 18 will have their records abstracted by study staff.
* Starting in the 13th month after PredicTB implementation (i.e., after the 12-month post-implementation period has ended), study staff will position themselves in the four study clinics for purposes of recruiting and enrolling adult patients submitting sputum for a new diagnosis of pulmonary TB. No exclusions will be made except for age (as above), and we will seek to enroll all consecutive patients until our target sample size (25 participants per clinic, total n = 100) has been reached.

Exclusion Criteria:

* Age < 15 years old

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3332 (Actual)
Dates: Start 2021-11-10 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2024-02-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David W Dowdy, MD/PHD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Makerere University, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baik Y, Musoke M, Twinamasiko A, Lamunu M, Nabacwa V, Sanyu A, Robsky KO, Sung J, Kityamuwesi A, Katamba A, Dowdy DW. Effectiveness and Implementation of a Clinical Risk Score for Early Diagnosis of Tuberculosis in Uganda: A Pragmatic, Clustered Randomization Clinical Trial. Ann Am Thorac Soc. 2025 Oct;22(10):1476-1483. doi: 10.1513/AnnalsATS.202404-422OC. PMID 40587503

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was initially conducted in eight primary health clinics (four clinics in the intervention arm and the other four clinics in the control arm). During the study, a total of three clinics (two in the intervention arm and one in the control arm) were replaced with other facilities of similar size and location for the remainder of the study period, resulting in 11 participating clinics.
Units Other Than Participants: Clinics
Groups:
- Score Intervention Arm: The PredicTB score will be implemented in this arm.
  PredicTB score: This is an easy-to-use clinical risk score designed to improve early management of tuberculosis in highly resource-constrained settings where same-day microbiological testing is unavailable. It consists of readily accessible demographic and clinical data and is scored from 1-10.
  We will train clinic staff in eight clinics (four study clinics and four comparison clinics) on the Ugandan standard of care for the diagnosis and treatment of TB. In addition, in the four study clinics, we will provide training on the PredicTB score.
Period: Overall Study
Arm/Group | Score Intervention Arm | Control Arm
Started | 1826; 6 Clinics | 1506; 5 Clinics
Completed | 1826; 6 Clinics | 1506; 5 Clinics
Not Completed | 0; 0 Clinics | 0; 0 Clinics

BASELINE CHARACTERISTICS:
Units Other Than Participants: Clinics
Groups:
- Total: Total of all reporting groups
Arm/Group | Score Intervention Arm | Control Arm | Total
Number analyzed (Participants) | 1826 | 1506 | 3332
Number analyzed (Clinics) | 6 | 5 | 11
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 36 [27 to 47] | 35 [27 to 47] | 36 [27 to 48]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One missing in sex at control arm
  Participants
    number analyzed (Participants) | 1826 | 1505 | 3331
    Female | 1077 | 834 | 1911
    Male | 749 | 671 | 1420
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0 | 0 | 0
    (all) |  |  | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Uganda | 1826 | 1506 | 3332
HIV status [Count of Participants; unit: Participants]
  Positive | 857 | 684 | 1541
  Negative | 760 | 741 | 1501
  Unknown/Missing | 209 | 81 | 290
Sputum specimen submitted [Count of Participants; unit: Participants] | 1348 | 1007 | 2355
Microbiologically confirmed TB [Count of Participants; unit: Participants] | 173 | 138 | 311

OUTCOME MEASURES:

1. Primary Outcome: Difference in 7-day Treatment Initiation From Pre-implementation to Post-implementation
Description: The percentage of participants with microbiologically confirmed TB who initiated treatment within 7 days during post-implementation 'minus' The percentage of participants with microbiologically confirmed TB who initiated treatment within 7 days during pre-implementation
Time Frame: Up to 12 months post intervention
Population: This outcome includes individuals who were diagnosed with tuberculosis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Score Intervention Arm | Control Arm
Number analyzed (Participants) | 1036 | 574
percentage of participants | 1 [-6 to 8] | -13 [-22 to -5]

2. Primary Outcome: Implementation: Percentage of Encountered Patients at Intervention Arm Who Initiated the Same-day Treatment Based on PredicTB Score as Indicated
Description: Percentage of patients who initiated same-day treatment divided by the number of patients who had a higher PredicTB score than the clinic-specific score of treatment threshold in the post-implementation period in intervention arm
Time Frame: Up to 12 months
Population: This outcome includes individuals who presented TB symptoms. This outcome is relevant to intervention arm only.
Measure: Number; unit: percentage of participants
Arm/Group | Score Intervention Arm | Control Arm
Number analyzed (Participants) | 229 | 0
percentage of participants | 46 |

3. Secondary Outcome: Incremental Cost-effectiveness of PredicTB
Description: (cost of implementing PredicTB - cost of standard of care)/(projected disability-adjusted life years (DALYs) in standard of care - projected DALYs with PredicTB)
Time Frame: Months 0 - 12
Population: Data was not collected.
Arm/Group | Score Intervention Arm | Control Arm
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Difference in TB Mortality From Pre-implementation to Post-implementation
Description: The percentage of participants with microbiologically confirmed TB who died of any cause in the post-implementation "minus" The percentage of participants with microbiologically confirmed TB who died of any cause in the pre-implementation
Time Frame: 12 Months
Population: This outcome includes individuals who were diagnosed with tuberculosis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Score Intervention Arm | Control Arm
Number analyzed (Participants) | 1036 | 574
percentage of participants | -1 [-4 to 1] | -1 [-6 to 5]

5. Secondary Outcome: Difference in Loss to Care From Pre-implementation To Post-implementation
Description: The percentage of participants with microbiologically confirmed TB who were lost to follow-up in the post-implementation "minus" The percentage of participants with microbiologically confirmed TB who were lost to follow-up in the pre-implementation
Time Frame: 12 Months
Population: This outcome includes individuals who were diagnosed with tuberculosis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Score Intervention Arm | Control Arm
Number analyzed (Participants) | 1036 | 574
percentage of participants | 1 [-3 to 2] | 1 [-5 to 3]

6. Secondary Outcome: Difference in Percentage of Participants With Microbiologically Confirmed TB
Description: Difference in the percentage of participants with microbiologically confirmed TB who initiated treatment within 7 days from post-implementation to pre-implementation at intervention arm "minus" Difference in the percentage of participants with microbiologically confirmed TB who initiated treatment within 7 days from post-implementation to pre-implementation at comparison arm
Time Frame: Up to 12 months post-implementation
Population: This outcome includes individuals who were diagnosed with tuberculosis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Score Intervention Arm | Control Arm
Number analyzed (Participants) | 1036 | 574
percentage of participants | 14 [10 to 19] | 0 [0 to 0]

7. Secondary Outcome: Reach: Percentage of Patients Who Were Administered (or Evaluated) by PredicTB Score
Description: Percentage of patients who were administered (or evaluated) by PredicTB score among those who presented presumptive TB symptoms at clinics in the post-implementation period in intervention arm
Time Frame: Up to 12 months
Population: This outcome includes individuals who presented TB symptoms. This outcome is relevant to intervention arm only.
Measure: Number; unit: percentage of participants
Arm/Group | Score Intervention Arm | Control Arm
Number analyzed (Participants) | 1826 | 0
percentage of participants | 66 |

8. Secondary Outcome: Adoption: Percentage of Providers Adopting PredicTB
Description: Percentage of providers using PredicTB in over 50% of encounters in which sputum is submitted for pulmonary TB diagnosis among those seeing >5 patients who submit sputum for diagnosis of pulmonary TB
Time Frame: Month 18
Population: This outcome analysis is relevant to intervention arm only. Per protocol, healthcare providers were not considered enrolled.
Measure: Number; unit: percentage of providers
Arm/Group | Score Intervention Arm | Control Arm
Number analyzed (Participants) | 17 | 0
percentage of providers | 100 |

9. Secondary Outcome: Maintenance: Change in Effectiveness Over Time in the Post-implementation Phase at Intervention Arm
Description: Percentage of participants with microbiologically confirmed TB who initiated treatment within seven days in the post-implementation phase at intervention arm "minus" Percentage of participants with microbiologically confirmed TB who initiated treatment within seven days in the post-implementation phase at intervention arm
Time Frame: Up to 12 months
Population: This outcome is relevant to intervention arm only
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Score Intervention Arm | Control Arm
Number analyzed (Participants) | 165 | 0
percentage of participants | -16 [-31 to 1] |

10. Secondary Outcome: Modeled Changes in 5-year Mortality With PredicTB
Description: Modeled hypothetical, expected changes in mortality at year 5, comparing simulations in which PredicTB is implemented to those in which PredicTB is not implemented, using a Markov state-transition model
Time Frame: Month 12
Population: Data was not collected.
Arm/Group | Score Intervention Arm | Control Arm
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: An average of 281 days
Description: Per Study Protocol, all-cause mortality and (serious and other than serious) adverse events were collected only from individuals who were diagnosed with tuberculosis during the post-implementation phase. Therefore, the number at risk is different from the number of participants with tuberculosis symptom presentation (the starting number of participants of the study).
Arm/Group | Score Intervention Arm | Control Arm
All-Cause Mortality (participants affected / at risk) | 12/316 | 17/211
Serious Adverse Events (participants affected / at risk) | 0/316 | 0/211
Other Adverse Events (participants affected / at risk) | 0/316 | 0/211

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-08-03): https://cdn.clinicaltrials.gov/large-docs/24/NCT05122624/Prot_SAP_000.pdf
  • Informed Consent Form (2021-05-21): https://cdn.clinicaltrials.gov/large-docs/24/NCT05122624/ICF_001.pdf